CLINICAL TRIAL: NCT05071144
Title: Advanced SPinal Innovations With Robotics and Enabling Technology Registry
Acronym: ASPIRE
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Pediatric Orthopaedic Society of North America (Other); Medtronic (Industry); Children's Hospital Colorado (Other); Hospital for Special Surgery, New York (Other); Children's Healthcare of Atlanta (Other); Rainbow Babies and Children's Hospital (Other); Dell Children's Medical Center of Central Texas (Other); Cedars-Sinai Medical Center (Other); Medical University of South Carolina Shawn Jenkins Children's Hospital (Other); St. Luke's Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Hedequist, Principal Investigator, Boston Children's Hospital
Other Study IDs: IRB-P00039760
Record Dates: First submitted 2021-09-07; First posted 2021-10-08 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Spine Deformity; Idiopathic Scoliosis; Adolescent Idiopathic Scoliosis; Spondylolisthesis; Congenital Scoliosis; Neuromuscular Scoliosis
Keywords: Pediatric; Spine; Surgery; Registry; Robotic; Navigation
MeSH Terms: conditions — Spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Spine Deformity Patients: Standard of care surgery using robotics coupled with navigation and/or patient-specific rods

SUMMARY:
Creation of a pediatric robotic spine surgery registry will allow for data collection and analysis on the coupled use of robotics and navigation, as well as patient-specific rods in pediatric spine deformity surgery across participating study institutions. Eventually, an educational and informative framework for this technology will be established.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a spine deformity
* Scheduled for surgery using robotics and navigation and/or patient-specific rods
* Up to and including 21 years of age
* Speak and read English or Spanish

Exclusion Criteria:

• None

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Study participants will be those receiving treatment for spinal deformity at one of the participating sites. Eligible patients will be identified from clinical databases of children undergoing surgery for spinal deformity.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
proportion of pedicle screws within 2 mm of cortical breach | Time of surgery
  The proportion of pedicle screws within 2 mm of cortical breach when assessed on intraoperative O-arm scans and postoperative CT scans (when applicable).

SECONDARY OUTCOMES:
radiation dose to patient and surgeon per screw | Time of surgery
  Radiation dose to patient and surgeon per screw based on the following imaging studies when performed: preoperative CT scan, intraoperative O-arm scans, and fluoroscopy.
Scoliosis Research Society (SRS-30) Questionnaire | Baseline, 6 Months, 1 Year, 2 Years, and 5 Years
  Questionnaires will be completed by both the patient and caregiver based on their appropriate diagnosis (i.e. idiopathic, congenital, spondylolisthesis, etc.).
Early Onset Scoliosis 24-Item Questionnaire (EOSQ-24) | Baseline, 6 Months, 1 Year, 2 Years, and 5 Years
  Questionnaires will be completed by both the patient and caregiver based on their appropriate diagnosis (i.e. idiopathic, congenital, spondylolisthesis, etc.).
Caregiver Priorities & Child Health Index of Life with Disabilities (CP Child) | Baseline, 6 Months, 1 Year, 2 Years, and 5 Years
  Questionnaires will be completed by both the patient and caregiver based on their appropriate diagnosis (i.e. idiopathic, congenital, spondylolisthesis, etc.).
Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Activity | Baseline, 6 Months, 1 Year, 2 Years, and 5 Years
  "Self-reported capability rather than actual performance of physical activities. This includes the functioning of one's upper extremities (dexterity), lower extremities (walking or mobility), and central regions (neck, back), as well as instrumental activities of daily living."
Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress - Anxiety | Baseline, 6 Months, 1 Year, 2 Years, and 5 Years
  "Fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness)."
Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress - Depressive Symptoms | Baseline, 6 Months, 1 Year, 2 Years, and 5 Years
  "Negative mood (sadness, guilt), views of self (self- criticism, worthlessness), and social cognition (loneliness, interpersonal alienation), as well as decreased positive affect and engagement (loss of interest, meaning, and purpose)."
Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function - Mobility | Baseline, 6 Months, 1 Year, 2 Years, and 5 Years
  "Activities of physical mobility such as getting out of bed or a chair to activities such as running."
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain - Interference | Baseline, 6 Months, 1 Year, 2 Years, and 5 Years
  "Consequences of pain on relevant aspects of one's life. This includes the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities."
Patient-Reported Outcomes Measurement Information System (PROMIS) Peer Relationships | Baseline, 6 Months, 1 Year, 2 Years, and 5 Years
  "Quality of relationships with friends and other acquaintances."
Operative time | Time of surgery
  Data collection on time related to robotics-navigation, including registration, screw planning, screw placement, and total time related to platform use defined as the beginning of registration to last screw placement.
Estimated blood loss (EBL) | Time of surgery
  EBL during surgery will be reported by the surgeon or extracted from surgical documentation.
Total operative cost | Time of surgery
  Capital expenses associated with the equipment and software, preoperative planning time, surgical time, and costs for revision surgery caused by screw malposition.
Improvement to spinopelvic alignment with PSR | Baseline, Predicted plan, 6 months, 1 year, 2 years, 5 years
  Spinopelvic alignment parameters including pelvic tilt, pelvic incidence, lumbar lordosis, thoracic kyphosis and sagittal vertical axis

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hedequist, MD, Principal Investigator — Boston Children's Hospital
Locations (10):
- United States (10):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - St. Louis Children's Hospital, St Louis, Missouri
  - Hospital for Special Surgery, New York, New York
  - Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Medical University of South Carolina Shawn Jenkins Children's Hospital, Charleston, South Carolina
  - Dell Children's Medical Center, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
The data for this study may also be sent to the Pediatric Spine Foundation Study Group (PSSG) and/or the HARMS Study Group in the future. The study data may be stored in PSSG for use in future research studies conducted by the members of PSSG. To help protect participant confidentiality, any data we send to these groups will not include their name or any other identifying information. Data will be tagged with a study ID.
Supporting Information: Study Protocol
Time Frame: The sharing timeline is dependent on study investigators and will be considered after enrollment closure.